CLINICAL TRIAL: NCT04686682
Title: A Phase I/IIa, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-8263 in Adult Patients With Advanced Malignant Tumors
Brief Title: A First-in-Human, JAB-8263 in Adult Patients With Advanced Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-8263-1002
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: NSCLC; SCLC; CRPC; ESCC; Ovarian Carcinoma; AML; MF; Malignant Tumor
Keywords: BET inhibitor; Bromodomain and Extra-terminal
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JAB-8263 Part1 (Experimental): Monotherapy, dose escalation
  Interventions: Drug: JAB-8263
- JAB-8263 Part 2 (Experimental): Monotherapy, dose expansion
  Interventions: Drug: JAB-8263

INTERVENTIONS:
Drug: JAB-8263 — Variable dose, orally Q2D with 28 days each cycle
  Arms: JAB-8263 Part1
Drug: JAB-8263 — RP2D dose, orally Q2D with 28 days each cycle
  Arms: JAB-8263 Part 2

SUMMARY:
This is a Phase 1/2a, first-in-human, open-label study of JAB-8263, this study has two parts: solid tumor dose escalation and expansion study and hematology tumor dose escalation and expansion study.

These two parts will determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D) and assess the DLT of JAB-8263 in treatment with patients with advanced solid tumors and hematology tumors separately. 30 subjects each will be enrolled.

DETAILED DESCRIPTION:
JAB-8263 is a small-molecule inhibitor of the highly conserved bromodomain pockets of the bromodomain and extraterminal (BET) proteins.

The objectives of this study are:

To determine the maximum-tolerated dose (MTD) and assess the dose-limiting toxicity (DLT) of JAB-8263 as a single agent to adult subjects with advanced malignant tumors. To assess the safety and tolerability of JAB-8263 To characterize the pharmacokinetic (PK) parameters and pharmacodynamics (PDc).To evaluate preliminary antitumor activity of JAB-8263

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following criteria in order to be included in the research study:

  1. Subject must be ≥18 years-of-age at the time of signature of the informed consent form (ICF).
  2. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
  3. Subjects with histologically or cytologically confirmed advanced solid tumors which have progressed despite standard therapy(ies), or are intolerant to standard therapy(ies), or have a tumor for which no standard therapy(ies) exists.
  4. Subjects with recurrent/refractory AML according to WHO 2016
  5. Subjects with life expectancy ≥3 months.
  6. Patients with solid tumor must have at least one measurable lesion as defined by RECIST v1.1.
  7. Patients who have sufficient baseline organ function.

Exclusion Criteria:

1. History (≤3 years) of cancer that is histologically distinct from the cancer under study.
2. Known serious allergy to investigational drug or excipients
3. Active brain or spinal metastases
4. History of pericarditis or Grade ≥2 pericardial effusion
5. History of interstitial lung disease.
6. History of Grade ≥2 active infections within 2 weeks
7. Known human immunodeficiency virus (HIV) infection
8. Seropositive for hepatitis B virus (HBV)
9. Seropositive for hepatitis C virus (HCV), or HCV-RNA viral levels are not detectable.
10. Any severe and/or uncontrolled medical conditions
11. History of myocardial infarction, unstable angina pectoris, coronary artery bypass graft, or cerebrovascular accident
12. Impaired cardiac function or clinically significant cardiac diseases
13. QTcF >470 msec at screening
14. History of medically significant thromboembolic events or bleeding diathesis
15. Unresolved Grade >1 toxicity
16. History of malignant biliary obstruction
17. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | Approximately 18 months
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with JAB-8263

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 18 months
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments
Area under the curve | Approximately 18 months
  Area under the plasma concentration time curve of JAB-8263
Cmax | Approximately 18 months
  Highest observed plasma concentration of JAB-8263
Tmax | Approximately 18 months
  Time of highest observed plasma concentration of JAB-8263
T1/2 | Approximately 18 months
  Half life of JAB-8263
Objective response rate ( ORR ) | Approximately 18 months
  For solid tumor study part, ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of response ( DOR ) | Approximately 18 months
  For solid tumor study part, DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Duration of response ( DCR ) | Approximately 18 months
  For solid tumor study part, DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD).
CR without minimal residual disease rate (CR MRD-) | Approximately 18 months
  hematology study part, CR MRD- is defined as proportion of participants with complete response without minimal residual disease.
Overall response rate | Approximately 18 months
  For hematology study part, Overall response rate is defined as proportion of participants with complete response(CR or CRi), partial remission(PR) or morphologic leukemia-free state(MLFS).
Event-free survival( EFS) | Approximately 18 months
  For hematology study part, EFS is defined for all patients with AML, measured from the date of entry into the study to the date of primary refractory disease, or relapse from CR, or Cri, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobio Pharmaceuticals, Study Director — Jacobio Pharmaceuticals
Locations (1):
- Tianjin, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No